CLINICAL TRIAL: NCT04623723
Title: Influence of Scaler Tip Design on Patients' Pain Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Nor Adinar Baharuddin, Associate Professor, University of Malaya
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 101269-5
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded (subject)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perio Slim (PS) (Sham Comparator): Supragingival scaling with a portable ultrasonic scaler device (EMS®) with PS (DS-016A, EMS® Piezon, Switzerland) scaler tip
  Interventions: Other: PS (DS-016A, EMS® Piezon, Switzerland) scaler tips. )
- Conventional scaler tip (Active Comparator): Supragingival scaling with a portable ultrasonic scaler device (EMS®) with conventional (FS-407, EMS® Piezon, Switzerland) scaler tip
  Interventions: Other: Conventional (FS-407, EMS® Piezon, Switzerland)

INTERVENTIONS:
Other: PS (DS-016A, EMS® Piezon, Switzerland) scaler tips. ) — Supragingival scaling with a portable ultrasonic scaler device (EMS®) with Piezon, Switzerland using PS (DS-016A, EMS® Piezon, Switzerland) scaler tips
  Arms: Perio Slim (PS)
Other: Conventional (FS-407, EMS® Piezon, Switzerland) — Supragingival scaling with a portable ultrasonic scaler device (EMS®) with Piezon, Switzerland using Conventional (FS-407, EMS® Piezon, Switzerland)
  Arms: Conventional scaler tip

SUMMARY:
Ultrasonic scalers have been shown effective in removing subgingival calculus. However, it may cause alteration to the tooth surface as well as discomfort to patients. Advances in scaler tip designs may reduce these effects. Limited studies have investigated the influence of scaler tip designs on tooth surface and patients' comfort. This study aimed to evaluate the influence of scaler tip designs on patients' pain perception.

DETAILED DESCRIPTION:
Scaling is a common procedure performed by general dental practitioners and dental specialists. Unfortunately, scaling has been associated with unpleasant dental treatment and to some extent, a painful experience (Berggren & Meynert, 1984). Studies also have demonstrated that scaling using ultrasonic scalers can cause tooth surface roughness and tooth substance loss (Jepsen et al., 2004; Kawashima et al., 2007). Rough tooth surface will increase retention of plaque and has been shown associated with early biofilm formation (Teughels et al., 2006). Subsequently, this would increase the risk for development and progression of periodontal disease. Whereas, tooth substance loss may lead to exposed dentinal tubules, and subsequently root sensitivity. Root sensitivity was reported to affect half of patients receiving periodontal therapy (Von Troil et al., 2002). This led to discomfort among patients and avoidance to dental treatment in future.

Advanced development in scaler tip designs has provided opportunities to deliver scaling treatment that is less aggressive to tooth surfaces and most importantly, to reduce the discomfort to patients. The design of the scaler tip has influenced the performance of ultrasonic scalers characterised by the displacement amplitude (Lea et al., 2003b). Displacement amplitude is the lateral movement of scaler tip that is thought to contribute to the aggressiveness of scaling procedure. Several studies have investigated the factors that may influence displacement amplitude, such as power setting and type of generator (Lea et al., 2003a), tip wear (Lea et al., 2006) and scaler tip designs (Lea et al., 2003a). However, to date, there were limited studies that investigated the effect of ultrasonic scaler tip design particularly slim and wide scaler tip on tooth surface roughness, tooth substance loss, and patients' pain perception.

In a clinical setting, if there were two treatment methods that provide similar levels of effectiveness but different levels of discomfort and damage to tooth surface patient will opt for the more comfortable and conservative method. Therefore, this study investigated the influence of scaler tip designs on tpatients' pain perception following scaling.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients aged 20-40 years who had anterior maxillary teeth from teeth #13 to #23.
* Diagnosed with chronic gingivitis and/or mild chronic periodontitis and presented with bleeding on probing (BOP) and minimal calculus from teeth #13 to #23

Exclusion Criteria:

* Smokers,
* Patients who had dentinal hypersensitivity, crowns, large restorations, non-vital teeth, acute dental infections or cervical lesions involving teeth #13 to #23.
* Patients who were on long-term non-steroidal anti-inflammatory drug therapy, undergoing orthodontic treatment or using removable partial dentures involving teeth from teeth #13 to #23

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-10-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Pain perception | 6 months
  Pain perception was assessed using the Visual Analogue Scale (VAS), which consists of a line numbered from 0 to 10. Scale '0' indicates no pain, whereas scale '10' indicates the worst possible pain. Participants were asked to score any number between these two ends that described the pain they experienced during treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berggren U, Meynert G. Dental fear and avoidance: causes, symptoms, and consequences. J Am Dent Assoc. 1984 Aug;109(2):247-51. doi: 10.14219/jada.archive.1984.0328. PMID 6590605
- [Result] Jepsen S, Ayna M, Hedderich J, Eberhard J. Significant influence of scaler tip design on root substance loss resulting from ultrasonic scaling: a laserprofilometric in vitro study. J Clin Periodontol. 2004 Nov;31(11):1003-6. doi: 10.1111/j.1600-051X.2004.00601.x. PMID 15491317
- [Result] Kawashima H, Sato S, Kishida M, Ito K. A comparison of root surface instrumentation using two piezoelectric ultrasonic scalers and a hand scaler in vivo. J Periodontal Res. 2007 Feb;42(1):90-5. doi: 10.1111/j.1600-0765.2006.00924.x. PMID 17214645
- [Result] Teughels W, Van Assche N, Sliepen I, Quirynen M. Effect of material characteristics and/or surface topography on biofilm development. Clin Oral Implants Res. 2006 Oct;17 Suppl 2:68-81. doi: 10.1111/j.1600-0501.2006.01353.x. PMID 16968383
- [Result] von Troil B, Needleman I, Sanz M. A systematic review of the prevalence of root sensitivity following periodontal therapy. J Clin Periodontol. 2002;29 Suppl 3:173-7; discussion 195-6. doi: 10.1034/j.1600-051x.29.s3.10.x. PMID 12787217
- [Result] Lea SC, Landini G, Walmsley AD. Displacement amplitude of ultrasonic scaler inserts. J Clin Periodontol. 2003 Jun;30(6):505-10. doi: 10.1034/j.1600-051x.2003.00012.x. PMID 12795788
- [Result] Lea SC, Landini G, Walmsley AD. Ultrasonic scaler tip performance under various load conditions. J Clin Periodontol. 2003 Oct;30(10):876-81. doi: 10.1034/j.1600-051x.2003.00395.x. PMID 14629574
- [Result] Lea SC, Landini G, Walmsley AD. The effect of wear on ultrasonic scaler tip displacement amplitude. J Clin Periodontol. 2006 Jan;33(1):37-41. doi: 10.1111/j.1600-051X.2005.00861.x. PMID 16367854
- [Derived] Abdul Hayei NA, Yahya NA, Safii SH, Saub R, Vaithilingam RD, Baharuddin NA. Influence of scaler tip design on root surface roughness, tooth substance loss and patients' pain perception: an in vitro and a randomised clinical trial. BMC Oral Health. 2021 Mar 31;21(1):169. doi: 10.1186/s12903-021-01540-0. PMID 33789646